CLINICAL TRIAL: NCT03737097
Title: Impact of Online Spaced Education on Long-term Retention of Knowledge About Fall Prevention by Patients With Multiple Sclerosis
Brief Title: Online Spaced Education to Improve Fall Prevention by Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HIAEfallMS
Record Dates: First submitted 2018-10-29; First posted 2018-11-09 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Education of Patients
Keywords: Fall; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Both arms will take place in the same period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Spaced Education (Experimental): The intervention cohort will participate in an online spaced education on fall prevention education developed for patients with multiple sclerosis.
  Interventions: Other: Online Spaced Education
- Brochure Education (Active Comparator): The control cohort will receive the fall prevention education in bolus through a Brochure developed by the National Multiple Sclerosis Society. The brochure was translated to portuguese and will be used in the study with authorization of the Society.
  Interventions: Other: Brochure Education

INTERVENTIONS:
Other: Online Spaced Education — Investigators created a set of fall prevention strategies for multiple sclerosis patients into an evidence-based form of online education, termed 'spaced education' (SE). Based upon two psychology research findings (the spacing and testing effects), spaced education has been shown in randomized trials to improve knowledge acquisition, boosts learning retention for up to two years, and durably improves changes in behavior.
  Arms: Online Spaced Education
Other: Brochure Education — The investigators translated and validated the Minimizing Your Risk of Falls A GUIDE FOR PEOPLE WITH MS brochure developed by the National Multiple Sclerosis Society. The control cohort will receive the main education model for patients that has been used in the past few years.
  Arms: Brochure Education

SUMMARY:
Multiple sclerosis (MS) is a chronic, progressive and neurodegenerative inflammatory disease that affects young adults. In many countries it has been described as the main cause of neurological incapacity in this age group. Due to the neurological impairment, patients with multiple sclerosis have a high incidence of fall. According to studies, MS patients fall three times more than general population. In the present study, the question to be answered is: education of individuals with MS on fall prevention using the method of online spaced education provides better retention of knowledge than the traditional method? This is a clinical trial to compare two methods of education of MS patients for prevention of fall. First stage: Development and validation of materials. Step two: Pilot questions with MS patients. Step three: Intervention and evaluation of outcome.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis diagnosis
* Accept to be part in the study
* Have valid e-mail address

Exclusion Criteria:

- Healthcare professionals;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in test scores between cohorts measured in weeks 1-24 | Months 1-6
  Test scores on fall prevention strategies tests in both cohorts will be registered and compared in weeks 1, 12 and 24

SECONDARY OUTCOMES:
Fall rate | Months 1-6
  Number of self-reported falls registered by the patients in both cohorts will be compared in weeks 1, 12 and 24
Adherence to fall prevention strategies | Months 1-6
  The study will apply the Falls Prevention Strategies Survey in both cohorts in weeks 1, 12 and 24. It is a self-report instrument addressing protective behaviors related to fall risk among adults with multiple sclerosis (MS) (eg, monitoring MS symptoms, wearing proper footwear, modifying activities). Response options reflect the frequency with which the respondent engages in the behavior (ie, never, sometimes, regularly)
Individuals satisfaction with the fall prevention education method | Months 3-6
  Individuals will be asked to evaluate their satisfaction with the method they were signed in the study by a five-point Likert scale (very dissatisfied, dissatisfied, neutral, satisfied, very satisfied). Answers will be compared between both cohorts in weeks 12 and 24.
Baseline knowledge levels of patients assessed via their initial responses to the questions | Month 1
  Previous knowledge about fall prevention strategies will be evaluated in week 1 in both cohorts and compared
Pre and post-test performances differences by age | Month 1-6
  Patient performance will be evaluated in both cohorts and compared by age in weeks 1, 12 and 24
Pre and post-test performances differences by gender | Month 1-6
  Patient performance will be evaluated in both cohorts and compared by gender in weeks 1, 12 and 24
Pre and post-test performances differences by history of falls | Months 1-6
  Patient performance in pre and post-tests will be evaluated in both cohorts and will be compared between fallers and non-fallers in the group and between the cohorts in weeks 1, 12 and 24. We will consider fallers the individuals, in both groups, that have at least one reported fall in the past six months in the enrollment in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar F Santos, PhD, Study Director — MD; Eliseth R Leão, PhD, Principal Investigator — Researcher
Locations (1):
- Sociedade Benef Israelitabras Hospital Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We do not plan to share IPD with other researchers